CLINICAL TRIAL: NCT04354714
Title: A Pilot Study of Ruxolitinib to Combat COVID-19
Brief Title: Ruxolitinib to Combat COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Could not make FDA required changes
Sponsor: Washington University School of Medicine (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-13-20-DiPersio
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ruxolitinib (Experimental): -Ruxolitinib is an oral medication that will be given twice daily (BID). Dosing on Days 1 through 3 will be 5 mg BID; dosing on Days 4 through 10 will be 10 mg BID.
  Interventions: Drug: Ruxolitinib; Procedure: Peripheral blood draw

INTERVENTIONS:
Drug: Ruxolitinib — For patients unable to swallow pills, a ruxolitinib suspension will be administered through a nasogastric/orogastric tube
  Other Names: Jakafi
Procedure: Peripheral blood draw — -Screening, Day 2, Day 4, Day 8, Day 15, and Day 29

SUMMARY:
The investigators hypothesize that JAK 1/2 inhibition with ruxolitinib, an FDA approved treatment for intermediate or high-risk myelofibrosis, could have a similar effect in patients with severe COVID-19, quelling the immune-hyperactivation, allowing for clearance of the virus and reversal of the disease manifestations.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of advanced COVID-19 as defined by both of the following:

  * A positive test for SARS-CoV-2 RNA detected by RT-PCR collected from the upper respiratory tract (nasopharyngeal and oropharyngeal swab) and, if possible, the lower respiratory tract (sputum, tracheal aspirate, or bronchoalveolar lavage), analyzed by a CLIA certified lab
  * Critical disease manifested by any of the following:

    * Chest imaging (CT or chest X-ray permitted) with ≥ 50% lung involvement
    * Respiratory failure requiring invasive mechanical ventilation or supplementary oxygen with FiO2 ≥ 50%
    * Shock (defined as mean arterial pressure ≤ 65 mmHg unresponsive to 25ml/kg isotonic intravenous fluid resuscitation and/or requiring vasopressor support
    * Cardiac dysfunction defined by:

      * New global systolic dysfunction with ejection fraction ≤ 40%
      * Takotsubo cardiomyopathy
      * New onset supraventricular or ventricular arrhythmias
      * Plasma troponin I ≥ 0.10 ng/mL in someone without previously documented troponin elevation beyond that level
      * Elevated plasma NT-proBNP in someone without documented prior elevation

        * If Age < 50, NT-proBNP > 450 pg/ml
        * If Age 50-74, NT-proBNP > 900 pg/ml
        * If Age ≥ 74, NT-proBNP > 1800 pg/ml
* Receipt of investigational or off-label agents for COVID-19 (prior or ongoing) does not exclude eligibility.
* Patients who have received autologous or allogeneic stem cell transplant are eligible at the discretion of the investigators.
* 18 years of age or older at the time of study registration
* Adequate hematologic function defined as:

  * absolute neutrophil count ≥ 1000/mm3
  * platelet count ≥ 50,000/mm3 without growth factor or transfusion support for 7 days prior to screening
* Creatinine clearance ≥ 15 mL/minute or receiving renal replacement therapy
* Women of childbearing potential (defined as women with regular menses, women with amenorrhea, women with irregular cycles, women using a contraceptive method that precludes withdrawal bleeding, or women who have had a tubal ligation) are required to have a negative pregnancy test and use two forms of acceptable contraception, including one barrier method, during participation in the study treatment period.
* Male patients (if engaging in reproductive sex with a women of childbearing potential) are required to use two forms of acceptable contraception, including one barrier method, during participation in the study and throughout the evaluation period.
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable)

Exclusion Criteria:

* Known allergy or intolerance to ruxolitinib or another JAK inhibitor.
* Known or suspected active viral (including HIV, hepatitis B, and hepatitis C), bacterial, mycobacterial, or fungal infection other than COVID-19. Virologic testing not required unless infection is suspected.
* Pregnant and/or breastfeeding.
* Any uncontrolled intercurrent illness that would put the patient at greater risk or limit compliance with study requirements in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Through 28 days

SECONDARY OUTCOMES:
Length of hospital stay | Through completion of follow-up (estimated to be 7 months)
Length of ICU stay | Through completion of follow-up (estimated to be 7 months)
Duration of ventilator use | Through completion of follow-up (estimated to be 7 months)
Duration of vasopressors use | Through completion of follow-up (estimated to be 7 months)
Duration on renal replacement therapy | Through completion of follow-up (estimated to be 7 months)
Viral kinetics as measured by virologic failure | Through completion of follow-up (estimated to be 7 months)
  -Defined as increase in viral load of >0.5 log on two consecutive days, or >1 log increase in one day, not in keeping with any baseline trend of rising viral loads during the pre-treatment viral testing
Number of adverse events as measured by CTCAE v. 5.0 | Through completion of follow-up (estimated to be 7 months)
Proportion of participants with detectable virus | Day 5
Proportion of participants with detectable virus | Day 10
Proportion of participants with detectable virus | Day 15
Proportion of participants with detectable virus | Day 29

CONTACTS AND LOCATIONS:
Overall Officials: John DiPersio, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu